CLINICAL TRIAL: NCT03803956
Title: Infrared Low-level Laser Therapy (Photobiomodulation Therapy) Before Intense Progressive Running Test of High-level Soccer Players: Effects on Functional, Muscle Damage, Inflammatory and Oxidative Stress Markers
Brief Title: Infrared Low-level Laser Therapy Before Intense Progressive Running Test of High-level Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Ernesto Cesar Pinto Leal Junior, Full professor, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 397774/2011
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Muscle; Fatigue, Heart; Skeletal Muscle Recovery
Keywords: Photobiomodulation therapy; Low-level laser therapy; Performance; Skeletal muscle recovery; High-level soccer players; Intense progressive running test
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: The volunteers who will receive active PBMT in the first stage of the study, will receive placebo PBMT in the second stage, while the volunteers that will receive placebo PBMT in the first stage, will receive active PBMT in the second stage of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The mode of intervention (active or placebo photobiomodulation) will be coded by an independent researcher. The randomization schedule will contain only codes (not the actual intervention). The output from the laser device is exactly the same from either the active or the placebo interventions. These features will guarantee that participants, therapists and outcomes assessor will be blinded to the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active PBMT (Active Comparator): Application of PBMT (Photobiomodulation Therapy) with a total dose of 850 Joules.
  Interventions: Device: Active PBMT
- Placebo PBMT (Placebo Comparator): Application of placebo PBMT (Photobiomodulation Therapy) without any dose (0 Joule).
  Interventions: Device: Placebo PBMT

INTERVENTIONS:
Device: Active PBMT — The PBMT will be performed using the dose of 10J per diode, previously determined by a previous study and power output of 100 mW per diode, also previously determined. PBMT will be performed at nine different sites of the knee extensor muscles, six different sites of the knee flexor muscles and two different sites of the plantar flex muscles. As the cluster will be 5 diodes and 17 different sites will be irradiated, a total of 85 points will be irradiated in each lower limb, a total of 850 J of energy. The active PBMT will be performed before a progressive running test.
  Arms: Active PBMT
Device: Placebo PBMT — The placebo PBMT will per performed using the dose of 0 J per diode. Placebo PBMT will be performed at nine different sites of the knee extensor muscles, six different sites of the knee flexor muscles and two different sites of the plantar flex muscles. As the cluster will be 5 diodes and 17 different sites will be irradiated, a total of 85 points will be irradiated in each lower limb, a total of 0 J of energy. To ensure blinding, the device emitted the same sound regardless of the programmed mode (active or placebo PBMT). The placebo PBMT will be performed before a progressive running test.
  Arms: Placebo PBMT

SUMMARY:
Photobiomodulation therapy (PBMT) has recently been used to alleviate postexercise muscle fatigue and enhance muscle recovery, demonstrating positive results. A previous study by the investigator's research group demonstrated the optimal dose and the optimal output power (100 mW) for an infrared wavelength (810 nm). However, the effects of optimized PBMT on performance and post-exercise recovery in high-level soccer players, to date have not been evaluated.

The present research project aims to evaluate the effects of PBMT (using low-level laser therapy) applied before a progressive running test on functional, muscle damage, inflammatory and oxidative stress markers in high-level soccer players.

DETAILED DESCRIPTION:
To achieve the proposed objective it will perform a randomized, crossover triple-blinded, placebo-controlled trial, with high-level soccer players as volunteers.

Twenty-two volunteers will be randomly allocated to two intervention groups: active or placebo PBMT before a progressive running test (ergospirometry test).

The blood samples for biochemical analysis will be obtained before and after a progressive running test, and another outcomes (functional) will be obtained during the test.

The data will be collected by a blind assessor. The statistical analysis will follow the intention-to-treat principles and data on functional analysis will be analyzed using the paired and two-tailed t-student test. Data on biochemical analysis will be analyzed using two-way ANOVA, followed by Bonferroni post hoc test.

The investigators will analyze: functional aspects (rates of oxygen uptake -VO2max (absolute and relative), aerobic and anaerobic threshold and time until exhaustion), muscle damage (creatine-kinase -CK and lactate dehydrogenase -LDH), inflammatory markers (IL-1β, IL-6 and TNF-α) and oxidative stress markers (Thiobarbituric acid -TBARS, catalase - CAT, superoxidedismutase - SOD and carbonylated proteins).

ELIGIBILITY:
Inclusion Criteria:

* High-level soccer players;
* Age between 18 and 35 years;
* Male gender;
* Minimum of 80% participation in team practice sessions;
* Agreement to participate through signed statement of informed consent.

Exclusion Criteria:

* History of musculoskeletal injury to hips or knees in previous 2 months;
* Use of pharmacological agents or nutritional supplements;
* Smokers and alcoholics;
* Occurrence of musculoskeletal injury during the trial;
* Any change in practice routine in relation to rest of the team during the trial.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Rates of oxygen uptake (VO2max). | Immediately after (1 minute) of ergospirometry test. Observation: the rates of oxygen uptake (relative and absolute) will be measured during the progressive running test.
  The rates of oxygen uptake will be measured by an ergospirometry test.

SECONDARY OUTCOMES:
Aerobic threshold. | Immediately after (1 minute) of ergospirometry test. Observation: the aerobic threshold will be measured during the progressive runThe aerobic and anaerobic threshold will be measured during the progressive running test.
  The aerobic threshold will be measured by an ergospirometry test.
Anaerobic threshold. | Immediately after (1 minute) of ergospirometry test (progressive running test). Observation: the aerobic threshold will be measured during the progressive running test.
  The anaerobic threshold will be measured by an ergospirometry test.
Activity of creatine kinase - CK. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Muscle damage will be measured by blood samples.
Activity of lactate dehydrogenase - LDH. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Muscle damage will be measured by blood samples.
Levels of interleukin 1 beta - IL-1b. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Inflammation will be measured by blood samples.
Levels of interleukin 6 - IL-6. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Inflammation will be measured by blood samples.
Levels of tumor necrosis factor alpha - TNF-a. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Inflammation will be measured by blood samples.
Levels of Thiobarbituric acid - TBARS | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Oxidative stress will be measured by blood samples.
Levels of carbonylated proteins. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Oxidative stress will be measured by blood samples.
Activity of catalase - CAT. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Oxidative stress will be measured by blood samples.
Activity of superoxidedismutase - SOD. | The blood samples will be collected 5 minutes after the ergospirometry test (progressive running test).
  Oxidative stress will be measured by blood samples.
Time until exhaustion. | Immediately after (1 minute) of ergospirometry test (progressive running test). Observation: the time until exhaustion will be measured during the progressive running test.
  The time until exhaustion will be measured by the software of ergospirometry system.

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Cesar Leal Junior, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Laboratory of Phototherapy and Innovative Technologies in Health, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tomazoni SS, Machado CDSM, De Marchi T, Casalechi HL, Bjordal JM, de Carvalho PTC, Leal-Junior ECP. Infrared Low-Level Laser Therapy (Photobiomodulation Therapy) before Intense Progressive Running Test of High-Level Soccer Players: Effects on Functional, Muscle Damage, Inflammatory, and Oxidative Stress Markers-A Randomized Controlled Trial. Oxid Med Cell Longev. 2019 Nov 16;2019:6239058. doi: 10.1155/2019/6239058. eCollection 2019. PMID 31827687